CLINICAL TRIAL: NCT04487951
Title: N-terminal Pro B-type Natriuretic Peptide and Vitamin D Levels as Prognostic Markers in COVID-19 Pneumonia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Collaborators: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Noha A. Radwan, Lecturer of Clinical and Chemical Pathology, Cairo University
Other Study IDs: 2020-7-1
Record Dates: First submitted 2020-07-24; First posted 2020-07-27 (Actual); Last update posted 2020-07-27 (Actual); Status verified 2020-07

CONDITIONS: COVID19 Pneumonia
Keywords: NT-pro-BNP; Vitamin D; COVID-19 Pneumonia; HPLC/UV Diode array
MeSH Terms: interventions — Vitamin D

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — serum samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Moderate: Moderate: moderate COVID -19 pneumonia
  Interventions: Other: Pro BNP , Vitamin D
- Severe: _severe COVID-19 pneumonia
  Interventions: Other: Pro BNP , Vitamin D

INTERVENTIONS:
Other: Pro BNP , Vitamin D — This study is designed to assess the difference between level of NT-pro-BNP, and Vitamin D in moderate cases who progressed to severe or critically ill category compared to those who did not.

SUMMARY:
This study is designed to assess the difference between level of NT-pro-BNP, and Vitmin D in moderate cases who progressed to severe or critically ill category compared to those who did not.

Assessment of any possible correlation between NT-pro-BNP and Vitamin D and the need for mechanical ventilation or mortality in COVID-19 infection.

DETAILED DESCRIPTION:
On 30 January 2020, World Health Organization (WHO) officially declared the COVID-19 epidemic as a public health emergency of international concern. An acute respiratory disease, caused by a novel coronavirus (SARS-CoV-2, previously known as 2019-nCoV), the coronavirus disease 2019 (COVID-19) has spread throughout China and received worldwide attention (Guo et al., 2020).

As an emerging acute respiratory infectious disease, COVID-19 primarily spreads through the respiratory tract, by droplets, respiratory secretions, and direct contact (Li et al., 2020). Based on current epidemiological investigation, the incubation period is 1-14 days, mostly 3-7 days and the COVID-19 is contagious during the latency period (Jin et al., 2020). The common clinical manifestations included fever (88.7%), cough (67.8%), fatigue (38.1%), sputum production (33.4%), shortness of breath (18.6%), sore throat (13.9%), and headache (13.6%) [16]. In addition, a part of patients manifested gastrointestinal symptoms, with diarrhea (3.8%) and vomiting (5.0%) (Guan et al., 2020).

B-type Natriuretic Peptide (BNP) is mainly synthesized and secreted by myocytes in the left ventricle (LV) as a response to myocytes stretched by pressure overload or volume expansion of the ventricle (Cao et al., 2019). In patients with Community Acquired Peumonia (CAP), NT-pro BNP levels are powerful predictors of adverse cardiac events. For patients with systemic inflammatory response syndrome (SIRS), Chen et al found that compared with non-SIRS patients, subjects with SIRS had a markedly higher level of B-type natriuretic peptide (BNP). Additionally, BNP level of more than 113 pg/mL was independent predictor of all-cause mortality in septic patients. Additionally, in 302 CAP patients, Christ-Crain et al confirmed that BNP levels increased with rising disease severity as classified by the pulmonary severity index (PSI) (p=0.01). Li et al confirmed that BNP could be used as a biomarker for evaluating the severity of CAP. They recommended BNP level of 299.0 pg/mL in predicting in-hospital mortality (sensitivity 67.5%, specificity 81.6%) (Zhang et al., 2016).

In respiratory system conditions, such as influenza, vitamin D has wide-ranging and fundamental roles, including through: gene transcription via COVID-19 relevant VDR (Vitamin D Receptor) pathways; wider immune function; and airway epithelial cell tight-junction function and integrity. Further, studies suggest vitamin D supplementation may be protective in respiratory conditions, the effect being highly significant in 'D' deficient persons. It is hypothesized by Watkins, 2020 and Grant et al., 2020 that vitamin D insufficiency may significantly compromise, respiratory immune response function, greatly increasing risk of COVID-19 severity and mortality (Brown and Sarkar, 2020).

Primary outcomes: This study is designed to assess the difference between level of NT-pro-BNP, and Vitmin D in moderate cases who progressed to severe or critically ill category compared to those who did not.

Secondary outcomes: Assessment of any possible correlation between NT-pro-BNP and Vitamin D and the need for mechanical ventilation or mortality in COVID-19 infection.

The study will be conducted on 100 COVID-19 confirmed patients Group (1): 50 mild to moderate cases (lung shadows without hypoxia and oxygen saturation >92%) who progressed to severe illness characterized by hypoxia necessitating oxygen therapy, or critical illness characterized by respiratory failure necessitating mechanical ventilation either invasive or non-invasive within their hospital stay.

Group (2): 50 mild to moderate cases who did not show clinical progression and were discharged.

ELIGIBILITY:
Inclusion Criteria:

* All cases will be diagnosed with COVID-19 by RT-PCR • Group (1) Critically ill patients: Respiratory Rate > 30/min SaO2 < 92% at room temperature Chest radiology showing more than 50% lesion or progressive lesion within 24 to 48 hours • Group (2) moderate cases: Patients has pneumonia manifestations on radiology associated with symptoms &/or leucopenia or lymphopenia.

Exclusion Criteria:

* Other causes of pneumonia other than infection with SARS-CoV-2.

  * Concomitant heart failure.
  * Hypoxic patients on hospital admission.
  * Arrhythmia.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study will be conducted on 100 COVID-19 confirmed patients Group (1): 50 mild to moderate cases (lung shadows without hypoxia and oxygen saturation >92%) who progressed to severe illness characterized by hypoxia necessitating oxygen therapy, or critical illness characterized by respiratory failure necessitating mechanical ventilation either invasive or non-invasive within their hospital stay.
  Group (2): 50 mild to moderate cases who did not show clinical progression and were discharged.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2020-11-01 (Estimated); Study Completion 2021-01-01 (Estimated)

PRIMARY OUTCOMES:
NT-pro-BNP and Vitamin D | 6 month
  level of NT-pro-BNP, and Vitamin D

SECONDARY OUTCOMES:
Assessment of any possible correlation between NT-pro-BNP and Vitamin D and the need for mechanical ventilation or mortality in COVID-19 infection | 6 month
  Assessment of any possible correlation between NT-pro-BNP and Vitamin D and the need for mechanical ventilation or mortality in COVID-19 infection

CONTACTS AND LOCATIONS:
Overall Officials: Akram Abdelbary, Prof., Principal Investigator — Cairo University
Locations (1):
- Kasr Alainy Cairo University, Cairo, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.